CLINICAL TRIAL: NCT07296302
Title: Randomized Clinical Trial Comparing Prophylactic Antibiotic Therapy and Placebo in Intraoral Alveolar Bone Grafting Procedures.
Brief Title: Antibiotic Prophylaxis Versus Placebo in Alveolar Bone Grafting: A Randomized Controlled Trial
Acronym: ABXGRAFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agnaldo Rocha de Souza Junior (Other)
Responsible Party: Sponsor-Investigator, Agnaldo Rocha de Souza Junior, Sponsor-Investigator, DDS, MSc, PhD, Universidade Estadual de Montes Claros
Organization: Universidade Estadual de Montes Claros (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARSJ-RCT-ABXGRAFT-01
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Alveolar Ridge Augmentation; Bone Grafting; Antibiotic Prophylaxis
Keywords: Ridge Preservation; Alveolar Bone Graft; Antibiotic Prophylaxis; Synthetic Bone Graft; Biphasic Calcium Phosphate
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: an amoxicillin group receiving 500 mg every 8 hours for 7 days and a placebo group receiving identical capsules. Both groups will undergo the same surgical protocol for alveolar bone grafting and will be followed at identical time points for clinical, radiographic, microbiological, and molecular assessments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcomes assessors will remain blinded to group allocation. Amoxicillin and placebo capsules are identical in appearance, packaging, and administration schedule. Randomization codes will be held by an independent researcher and will only be revealed after completion of all data collection and primary analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amoxicillin Prophylaxis Group (Active Comparator): Amoxicillin 500 mg 1 hour before surgery, followed by 500 mg every 8 hours for 7 days. In case of penicillin allergy, azithromycin 500 mg 1 hour before surgery followed by 500 mg once daily for 3 days.
  Interventions: Drug: Amoxicillin 500 mg (prophylactic regimen)
- Placebo Group (Placebo Comparator): Placebo capsules identical in appearance to the active medication. Dosing schedule matches the amoxicillin regimen: one capsule administered 1 hour preoperatively, followed by capsules every 8 hours for 7 days. For participants with documented penicillin allergy, placebo capsules will follow the azithromycin schedule (one dose preoperatively and one capsule daily for 3 days).
  Interventions: Drug: Placebo Capsule (matched dosing schedule)

INTERVENTIONS:
Drug: Amoxicillin 500 mg (prophylactic regimen) — Amoxicillin 500 mg administered 1 hour before surgery, followed by 500 mg every 8 hours for 7 days. Participants with documented penicillin allergy will receive azithromycin 500 mg 1 hour before surgery, followed by 500 mg once daily for 3 days.
  Arms: Amoxicillin Prophylaxis Group
Drug: Placebo Capsule (matched dosing schedule) — Participants will receive placebo capsules identical in appearance to the active medication, containing no active drug. One placebo capsule will be administered 1 hour before surgery, followed by placebo capsules every 8 hours for 7 days, matching the amoxicillin dosing schedule. Participants with documented penicillin allergy randomized to the placebo group will receive placebo capsules matching the azithromycin schedule (one dose preoperatively and one capsule daily for 3 days).
  Arms: Placebo Group

SUMMARY:
Tooth extraction sites often require alveolar bone grafting to preserve ridge dimensions and improve conditions for future implant placement. Although systemic antibiotic prophylaxis is commonly prescribed after grafting procedures, there is limited evidence supporting its necessity in healthy patients undergoing intraoral bone grafting. This randomized, double-blind, placebo-controlled clinical trial aims to compare the effects of prophylactic amoxicillin versus placebo on postoperative outcomes in alveolar bone graft procedures using Plenum® Oss HP biomaterial, a synthetic biphasic bioceramic composed of hydroxyapatite and beta-tricalcium phosphate (HA/β-TCP; 70:30 ratio).

Participants will be randomly assigned to receive either amoxicillin 500 mg every 8 hours for 7 days or a matching placebo. Clinical parameters, postoperative complications, and patient-reported outcomes will be assessed. The study seeks to determine whether antibiotic prophylaxis provides measurable clinical benefits or whether placebo yields comparable results, contributing to more rational antibiotic use and supporting antimicrobial stewardship in oral surgery.

DETAILED DESCRIPTION:
Alveolar bone grafting plays a central role in modern oral rehabilitation by preserving vertical and horizontal dimensions of the alveolar ridge following tooth extraction. The procedure is fundamental for optimizing future implant placement, reducing the need for additional regenerative surgeries, and improving long-term functional and esthetic outcomes. Despite its widespread use, postoperative management varies substantially among clinicians, particularly concerning the prescription of systemic antibiotic prophylaxis. Although antibiotics are often used empirically to prevent postoperative infection and graft failure, current scientific evidence remains inconclusive regarding their real benefit in healthy patients undergoing intraoral grafting under controlled aseptic conditions.

Antibiotic overprescription has important implications. Globally, antibiotic resistance is recognized as one of the most serious public health threats. Misuse of antibiotics in dentistry contributes significantly to this problem, especially when they are prescribed in situations where clinical benefit has not been firmly established. Additionally, unnecessary antibiotic use exposes patients to risks of adverse reactions, gastrointestinal disturbances, allergies, drug interactions, and increased treatment costs. In the specific context of alveolar bone grafts, the low incidence of postoperative infections reported in the literature raises questions about whether routine antibiotic prophylaxis is truly necessary.

This randomized, double-blind, placebo-controlled clinical trial was designed to rigorously evaluate whether postoperative amoxicillin provides measurable clinical, microbiological, or regenerative benefits compared with placebo in patients undergoing alveolar bone grafting using Plenum® OssHP, a synthetic biphasic bioceramic composed of hydroxyapatite and beta-tricalcium phosphate (HA/β-TCP; 70:30 ratio). The biomaterial is used in regenerative dentistry due to its osteoconductive properties and long-term volumetric stability. Its predictable behavior offers an ideal experimental environment to assess whether antibiotics influence early healing, infection rates, or the quality of regenerated bone.

Participants aged 18 years and older who require alveolar ridge preservation or augmentation with Plenum® Oss HP following tooth extraction will be recruited and screened according to the protocol approved by the Research Ethics Committee. After signing informed consent, eligible subjects will be randomly assigned in a 1:1 ratio to either the antibiotic group or the placebo group. Randomization will be stratified to reduce selection bias, and both participants and investigators will remain blinded throughout the study period. Individuals in the intervention group will receive amoxicillin 500 mg every 8 hours for 7 days, whereas the placebo group will receive identical capsules without active drug.

Surgical procedures will follow a standardized protocol, including atraumatic extraction when applicable, careful debridement of the alveolus, biomaterial placement, and tension-free flap closure. Postoperative care instructions and rescue medication protocols will be identical for all participants. Follow-up evaluations will occur at 7, 14, and 30 days, and again at 6 months during the re-entry procedure, allowing for multiple types of outcome assessment.

A comprehensive set of clinical, radiographic, histological, microbiological, proteomic, and metabolomic outcomes will be evaluated to understand the biological and clinical consequences of antibiotic use. The primary outcome is the incidence of postoperative infection at 7, 14, and 30 days. Infection will be clinically defined based on established diagnostic criteria including erythema, purulence, fever, increased pain, and delayed wound healing.

The secondary outcomes encompass a multidimensional assessment of healing. Radiographically, cone-beam computed tomography (CBCT) imaging will be obtained at baseline and at 6 months to evaluate bone volume gain, density, and mineralization patterns within the grafted region. These measurements provide insight into the structural maturation of the regenerated bone and allow quantitative comparison between groups.

Histomorphometric analysis will be performed using standardized biopsies collected at the time of implant placement or re-entry surgery. Samples will be processed and stained to quantify percentages of newly formed bone, residual biomaterial particles, and connective tissue. These indicators offer a precise understanding of the regenerative dynamics and the quality of bone formation influenced-or not-by antibiotic exposure.

Microbiological analysis will be carried out using sterile endodontic paper points placed in the surgical site at 7 and 14 days. Bacterial load will be quantified using established molecular or culture-based methods, enabling assessment of whether antibiotics modify early colonization patterns or microbial composition.

Beyond these measures, this study includes an innovative component: proteomic and metabolomic profiling of bone biopsy specimens. These high-throughput analyses provide a molecular-level understanding of tissue remodeling, inflammation, cellular metabolism, and bone regeneration pathways. Differences in protein expression profiles or metabolic signatures between antibiotic and placebo groups may reveal subtle biological effects not detectable through clinical or radiographic evaluation alone. This integrative biological approach may help identify biomarkers associated with bone healing and clarify mechanisms through which antibiotics could influence regenerative processes.

Patient-reported outcomes such as pain intensity, swelling, functional limitation, and overall treatment satisfaction will also be systematically recorded. Adverse events, including allergic reactions, gastrointestinal symptoms, or other complications, will be monitored to evaluate safety. By combining traditional clinical endpoints with advanced biological and imaging techniques, the study offers a comprehensive evaluation of healing trajectories following alveolar bone grafting.

The overarching goal of this trial is to determine whether postoperative antibiotic prophylaxis provides significant advantages over placebo in terms of infection control, bone regeneration quality, or patient comfort. If no measurable benefit is identified, the findings will support a reduction in unnecessary antibiotic use in dental regenerative procedures, contributing to antimicrobial stewardship and promoting safer, evidence-based clinical practice. Conversely, if antibiotics demonstrate clear advantages, their use can be better justified and applied selectively to patients who stand to benefit most.

Ultimately, this study is expected to generate high-quality evidence to inform clinical guidelines and optimize postoperative care in alveolar ridge preservation and augmentation procedures. By addressing an important knowledge gap, the trial seeks to improve patient safety, refine regenerative protocols, and contribute to global efforts against antibiotic overuse.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.

Generally healthy individuals classified as American Society of Anesthesiologists (ASA) physical status I or II ( ASA I or ASA II).

Indication for tooth extraction followed by alveolar bone grafting in a fresh socket.

Absence of active infection at the surgical site.

Willingness to take amoxicillin or, in cases of β-lactam antibiotic allergy, azithromycin.

No use of antibiotics in the previous 30 days.

Agreement to participate and signature of the informed consent form (ICF).

Exclusion Criteria:

* Presence of uncontrolled systemic diseases or chronic use of immunosuppressive medications.

Pregnancy or breastfeeding.

Severe liver disease.

Smoking more than 10 cigarettes per day.

Known allergy to macrolides (azithromycin).

Prior use of antibiotics within the last 30 days.

Concomitant use of medications with known risk of QT interval prolongation.

Signs of acute infection at the extraction site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative infection | 7, 14, and 30 days post-procedure
  Incidence of postoperative infection at 7, 14, and 30 days after alveolar bone grafting, assessed through clinical parameters including local pain, edema, purulent discharge, erythema, wound dehiscence, fever, and need for additional antibiotic therapy. Diagnosis will follow predefined clinical criteria.

SECONDARY OUTCOMES:
Volumetric bone formation and mineral density assessed by CBCT | Baseline and 6 months
  Volumetric bone gain and mineral density will be evaluated using cone-beam computed tomography (CBCT) scans performed at baseline and 6 months post-grafting. Standardized 3D segmentation will be applied to quantify bone formation and density changes within the grafted area.
Histomorphometric characteristics of regenerated bone | 6 months
  Histomorphometric assessment of bone biopsies collected at implant site reopening. Parameters include percentage of vital bone, residual graft particles, connective tissue, and inflammatory infiltrate.
Bacterial load at grafted sites | 7 and 14 days
  Bacterial load will be quantified from paper point samples collected at postoperative days 7 and 14. Quantification will include total bacterial burden and specific pathogens associated with postoperative infections.
Proteomic and metabolomic profile of regenerated bone tissue | 6 months
  Proteomic and metabolomic profiling will be performed on bone biopsy specimens to identify molecular pathways associated with healing, infection, inflammation, and graft integration.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual de Montes Claros - Unimontes, Montes Claros, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No